CLINICAL TRIAL: NCT03404219
Title: Enhancing Social Functioning in Schizophrenia Through Scalable Mobile Technology
Brief Title: Motivation and Skills Support (MASS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: San Francisco State University (Other)
Responsible Party: Principal Investigator, Daniel Fulford, Assistant Professor, Occupational Therapy and Rehabiltiation Sciences, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R21MH111501-01 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Mobile intervention (i.e., Ecological momentary intervention [EMI]) addressing social motivation and social skills. Twice daily notifications sent to deliver EMI content. Social goal reminders and steps provided to support goal attainment. Social Skills Training content delivered via brief video clips.
  Interventions: Behavioral: Motivation and Skills Support (MASS)

INTERVENTIONS:
Behavioral: Motivation and Skills Support (MASS) — Mobile phone-based application to support social skills and social motivation

SUMMARY:
Social impairment contributes to more severe symptoms, higher rates of hospitalization, and increased disability in persons with schizophrenia. In this study the investigators will develop a smartphone application and test its impact on improving real-world social functioning in persons with schizophrenia. Findings from this study will allow researchers and clinicians to better understand ways to improve social skills and social motivation, two common problems in the daily lives of persons with schizophrenia. The investigators hope this mobile phone-based support application will ultimately contribute to increased access to effective treatments for social functioning in this population.

DETAILED DESCRIPTION:
This project will involve an examination of the impact of a mobile intervention to improve social functioning in schizophrenia using an evidence-based treatment framework to target deficits in social skills and social motivation. Social impairment is a key characteristic of schizophrenia, present prior to onset and predictive of long-term course. The approach of the current project is to use Ecological Momentary Intervention (EMI), administered by mobile phone, to integrate features from social skills training (SST; an evidence-based treatment for schizophrenia) with social motivation support to improve social functioning. Aim 1 of the project will involve iterative development of the mobile application, using expert panel input and conducting usability testing to inform intervention content and approach. As an exploratory aim, social sensing technology (e.g., GPS and automated conversation detection) will be implemented to test the promise of this technology in identifying and intervening in social isolation. In Aim 2, 30 persons with schizophrenia will use the application over a 2-month period (data collection will occur across 2 sites). The investigators will test the impact of the application on social motivation (EMA reports of social anticipatory pleasure and presence of social interaction) across the intervention period. Investigators will also examine the impact on social functioning, measured with standard clinician-administered assessments, from baseline to 90-day follow-up. Additional clinical, neurocognitive, and social cognitive assessments will be gathered on study participants to identify potential moderators of outcome and predictors of application usability. This study will result in a better understanding of the feasibility and initial impact of a scalable intervention designed to support lasting, sustainable improvements in social functioning in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

•All participants with schizophrenia or schizoaffective disorder (identified either by self-report and confirmatory chart diagnosis, or by using the Structured Clinical Interview for DSM-5 [SCID-5]) will be in good general physical health, between 18 and 65 years old (as to not confound developmental issues with our focus), and fluent in English. Subjects do not need to have a significant other in order to participate in the study.

Exclusion Criteria:

•All participants with a current (past 6 months) substance use disorder, which will be determined by administration of the SCID-5, and self-reported current suicidal ideation with intent and/or a plan (assessed using attached instrument; i.e., "High" risk) or diagnosis of a neurological disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fulford, PhD, Principal Investigator — CRC BU Univeristy
Locations (2):
- United States (2):
  - San Francisco State University, San Francisco, California
  - Boston University, Boston, Massachusetts

REFERENCES:
- [Derived] Fulford D, Gard DE, Mueser KT, Mote J, Gill K, Leung L, Mow J. Preliminary Outcomes of an Ecological Momentary Intervention for Social Functioning in Schizophrenia: Pre-Post Study of the Motivation and Skills Support App. JMIR Ment Health. 2021 Jun 15;8(6):e27475. doi: 10.2196/27475. PMID 34128812

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 73 potential participants completed initial phone screen. 25 did not meet inclusion criteria based on age, neurological disorder status, recent hospitalization status, legal guardian status, or diagnosis. 48 participants were further screened. 10 of those participants did not meet inclusion criteria for diagnosis or substance use disorder status. 6 additional participants never initiated the intervention.
Groups:
- Intervention Group: All participants were assigned to this group and received the intervention.
Period: Overall Study
Arm/Group | Intervention Group
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Age, Continuous [Mean (Full Range); unit: years] | 46.097 [22 to 65]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 14
  Gender: Male | 16
  Gender: Unknown | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 14
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes in Social Functioning as Measured by the Social Functioning Scale (SFS)
Description: The Social Functioning Scale (SFS; Birchwood, Smith, Cochrane, Wetton, and Copestake, 1990) is a validated measure of social functioning commonly used in schizophrenia research studies. This clinician-administered measure consists of 7 sub-scales where higher scores indicate better social functioning: Social Engagement/Withdrawal (7 items. Score range: 0-15), Interpersonal (5 items. Score range: 0-30), Prosocial (5 items. Score range: 0-66), Recreation (23 items. Score range: 0-48), Independence - competence (15 items. Score range: 0-39), Independence - performance (13 items. Score range: 0-39), and Employment (13 items. Score range is 0-6 if the participant is unemployed and 7-10 if the participant is employed). The total score is the sum of the 7 sub-scales (Possible range of 0-247) and higher scores indicate better functioning. The investigators will examine the difference in total score from baseline (study entry) to follow-up (3 months after study termination).
Time Frame: Baseline (study entry) and follow-up (3 months post-intervention)
Population: Participants with schizophrenia or schizoaffective disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
score on a scale | 108.00 (7.13)
Statistical Analysis 1: Comparison: Intervention Group; Single arm; Test type: Other — Single group pre-post, follow-up; p = 0.09, General Linear Model (repeated measures); Mean Difference (Final Values) = 2.56

2. Primary Outcome: Changes in Social Engagement as Measured by the Quality of Life Scale (QLS) - Interpersonal Relations Subscale.
Description: The Heinrich Quality of Life Scale - Interpersonal Relations subscale (Heinrichs, Hanlon, & Carpenter, 1984) is a validated measure of social engagement used in studies of schizophrenia. This clinician-administered measure consists of 8 items that address different facets of social engagement (e.g., social network, acquaintances, intimate relationships, social withdrawal). Possible scores range from 0-48 with higher scores indicating better outcomes. The investigators will administer this measure at baseline (study entry) and follow-up (3 months post-intervention).
Time Frame: Baseline (study entry) and follow-up (3 months post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
score on a scale | 2.60 (1.36)

3. Secondary Outcome: Changes in Experience-Sampling-Based Self-Reports of Social Appraisals
Description: The investigators will ask participants to report on positive social appraisals (unpublished measure) of recent interactions 2 times per day over the 2-month intervention period. Specific items and response options are the following:
  1. "How well do you think you communicated in those conversations?" (from 1 [I did not communicate well at all] to 4 [I communicated very well])
  2. "To what extent were those interactions worth the effort?" (from 1 [not worth the effort at all] to 4 [definitely worth the effort])
  3. "What do you think other people thought of you in those conversations?" with response options ranging from 1 [very unlikable] to 4 [very likable]) We will average scores on the above items across all available time points (total possible time points = 120) to form a composite variable representing social appraisals. Higher scores represent more positive appraisals. Investigators will examine changes in appraisals over the intervention.
Time Frame: 2 times per day for 2 months (intervention period).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 31
score on a scale | 1.35 (0.64)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the full course of the study (total frame = 5 months).
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03404219/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT03404219/ICF_001.pdf